CLINICAL TRIAL: NCT01622062
Title: Verorab® Immunogenicity and Safety After a One-week, 4-site, Intradermal (ID) Post-exposure Prophylaxis Regimen (4-4-4-0-0) Followed by a One-visit, 4-site, ID Booster at Five Years
Brief Title: Immunogenicity and Safety of Verorab® in a "One-week" Intradermal Post-exposure Prophylaxis Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAB40; U1111-1122-2546 (Other: WHO)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Rabies
Keywords: Rabies; Verorab®; Favirab®
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Patients with WHO Category II exposure receive PEP with PVRV using "one-week, 4-site" (4-4-4-0-0) ID vaccination regimen, and a "single-visit, 4-site" booster vaccination with PVRV 5 years later
  Interventions: Biological: PVRV
- Group 2 (Experimental): Patients with WHO Category III exposure receive PEP with PVRV using "one-week, 4-site" (4-4-4-0-0) ID vaccination regimen and pERIG Favirab®, and a "single-visit, 4-site" booster vaccination with PVRV 5 years later
  Interventions: Biological: PVRV and pERIG Favirab®
- Group 3 (Active Comparator): Patients with WHO Category III exposure receive PEP with PVRV using the updated 2-site TRC (2-2-2-0-2) ID vaccination regimen and pERIG Favirab®, and a "single-visit, 4-site" booster vaccination with PVRV 5 years later
  Interventions: Biological: PVRV and pERIG Favirab®

INTERVENTIONS:
Biological: PVRV — 0.1 mL, 4 site 'one week' (4-4-4-0-0) administered intradermally
  Other Names: VERORAB®
  Arms: Group 1
Biological: PVRV and pERIG Favirab® — 0.1 mL of vaccine administered intradermally in 4 site 'one week' (4-4-4-0-0) regimen, and pERIG Favirab® (volume to be calculated according to the patient' body weight) infiltrated into and around wound(s)
  Other Names: VERORAB®; pERIG Favirab®
  Arms: Group 2
Biological: PVRV and pERIG Favirab® — 0.1 mL of vaccine administered intradermally in 2-site TRC (2-2-2-0-2) regimen, and pERIG Favirab® (volume to be calculated according to the patient' body weight) infiltrated into and around wound(s)
  Other Names: VERORAB®; pERIG Favirab®
  Arms: Group 3

SUMMARY:
The purpose of this study is to assess the 4-site "one-week" post-exposure prophylaxis (PEP) regimen as a possible alternative to the 2-site updated Thai Red Cross (TRC) PEP regimen.

Primary objective:

* To demonstrate that PEP using the new "one-week, 4-site" (4-4-4-0-0) intradermal (ID) vaccination regimen is non-inferior to PEP using the updated TRC (2-2-2-0-2) ID vaccination regimen.

Secondary objectives:

* Primary immunization: To describe the immune response in each group at Day 0, Day 14 and Day 90.
* Antibody persistence: To describe rabies virus-neutralizing antibody persistence during the 5 years after completion of PEP in each group.
* Booster vaccination: To describe the immune response induced by a single-visit 4-site intradermal booster vaccination in each group at Year 5.
* Safety: To describe the safety profile of each group after the primary and booster vaccinations.

DETAILED DESCRIPTION:
Participants with WHO Category II exposure will receive PEP, using "one-week, 4-site" ID vaccination regimen. Participants with WHO Category III exposure will receive PEP, using "one-week, 4-site" (4-4-4-0-0) ID vaccination regimen and pERIG Favirab® or using the updated 2-site TRC (2-2-2-0-2) ID vaccination regimen and pERIG Favirab®. All participants will receive a "single-visit, 4-site" booster vaccination five years later.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* Patient aged ≤50 years, with WHO category II or III contacts happened within 48 hours before appearance at site.

For adults:

* Informed consent form has been signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.

For children:

* For children under 18 years of age, informed consent form has been signed and dated by the parent(s) or another legally acceptable representative.
* For children under 18 years, assent form or informed consent form has been signed and dated by the appropriate age-range patient, according to country specific institution requirement as detailed in each country specific assent form or informed consent form.
* Patient and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

For all patients:

* Receipt of chloroquine or other medications used for malaria chemoprophylaxis, with or without other anti-malarial treatment, for more than 4 weeks (duration of anti-malarial course) and part of the treatment received within the 2 weeks before vaccination.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial immunization
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination, except for influenza vaccination and tetanus immunization (related only to current animal bite exposure
* Planned receipt of any vaccine in the 4 weeks following the trial primary and booster vaccination
* Previous immunization against rabies at any time in the past with either the trial vaccine and immunoglobulin or another rabies immunobiological product (in pre-or post-exposure regimen)
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus
* Patient with clinical signs of encephalitis
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator
* Febrile illness (temperature ≥38.0°C) or moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination
* Prior history of mammal animal bite within the past 5 years.

For infants or toddlers :

* Known personal or maternal seropositivity for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus, as reported by the parent/guardian
* Prior history of seizures .

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2012-06-29 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with seroconversion on Day 14 | Day 14 post vaccination
  Seroconversion is defined as rabies virus neutralizing antibody titers ≥ 0.5 IU/mL

SECONDARY OUTCOMES:
Percentage of participants with seroconversion before and after primary vaccination | Day 0, Day 14, Day 90
  Seroconversion is defined as rabies virus neutralizing antibody titers ≥ 0.5 IU/mL
Percentage of participants with seroconversion after primary vaccination (antibody persistence) | Year 1 to Year 5
  Seroconversion is defined as rabies virus neutralizing antibody titers ≥ 0.5 IU/mL
Percentage of participants with seroconversion after booster vaccination | Year 5 + 11 days
  Seroconversion is defined as rabies virus neutralizing antibody titers ≥ 0.5 IU/mL
Geometric mean titers (GMTs) before and after primary vaccination | Day 0, Day 14, Day 90
  Titers of rabies virus-neutralizing antibodies were assessed by the rapid fluorescent focus inhibition test
GMTs after primary vaccination (antibody persistence) | Year 1 to Year 5
  Titers of rabies virus-neutralizing antibodies were assessed by the rapid fluorescent focus inhibition test
GMTs after booster vaccination | Year 5 + 11 days
  Titers of rabies virus-neutralizing antibodies were assessed by the rapid fluorescent focus inhibition test
Number of participants reporting solicited injection site reactions following primary and booster vaccination | 7 days after each and any injection
  Solicited injection site reactions are tenderness (for participants aged ≤ 23 months), pain (for participants aged ≥ 2 years), redness and swelling (for all participants)
Number of participants reporting solicited systemic reactions following primary and booster vaccination | From Day 0 up to 7 days after injection 3, and 7 days after subsequent injections
  Solicited systemic reactions are Fever, Vomiting, Crying abnormal, Drowsiness, Appetite lost, and Irritability for participants aged ≤ 23 months and Fever (Temperature), Headache, Malaise, and Myalgia for participants aged ≥ 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Quiambao BP, Ambas C, Diego S, Bosch Castells V, Korejwo J, Petit C, Houillon G. Intradermal post-exposure rabies vaccination with purified Vero cell rabies vaccine: Comparison of a one-week, 4-site regimen versus updated Thai Red Cross regimen in a randomized non-inferiority trial in the Philippines. Vaccine. 2019 Apr 10;37(16):2268-2277. doi: 10.1016/j.vaccine.2019.02.083. Epub 2019 Mar 16. PMID 30890382
- See also: Related Info — http://www.sanofipasteur.com